CLINICAL TRIAL: NCT06843954
Title: Impact of Vascular Endothelial Growth Factor Gene Polymorphisms on Bevacizumab Efficacy in a Sample of Iraqi Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mohammed Mahmood Mohammed (Other)
Responsible Party: Sponsor-Investigator, Mohammed Mahmood Mohammed, Clinical associated professor, Al-Mustansiriyah University
Organization: Al-Mustansiriyah University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 106-38
Record Dates: First submitted 2024-08-23; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with mCRC and received bevacizumab (7.5mg/kg every 21 day) in association with combined regimen standard chemotherapy (FOLFOX, FOLFIRI, XELOX), at the end of the study NLR and PLR data were collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bevacizumab Group (Experimental): Patients diagnosed with mCRC and received bevacizumab (7.5mg/kg every 21 day) in association with combined regimen standard chemotherapy (FOLFOX, FOLFIRI, XELOX)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — bevacizumab (7.5mg/kg every 21 days) for minimum of 3 cycles

SUMMARY:
This study will be a prospective one conducted within a time frame between September 2022 and April 2023. One hundred adult patients already diagnosed with CRC and received bevacizumab and chemotherapy consisting of fluorouracil and leucovorin or capecitabine in combination with either oxaliplatin (FOLFOX or XELOX) or irinotecan (FOLFIRI or XELIRI). Three to six cycles will be given, and to explore the response to treatment, the Response Evaluation Criteria in Solid Tumors (RECIST) will be used to assess the response.

DETAILED DESCRIPTION:
This study will be a prospective one conducted within a time frame between September 2022 and April 2023. One hundred adult patients already diagnosed with CRC and received bevacizumab and chemotherapy consisting of fluorouracil and leucovorin or capecitabine in combination with either oxaliplatin (FOLFOX or XELOX) or irinotecan (FOLFIRI or XELIRI). Three to six cycles will be given, and to explore the response to treatment, the Response Evaluation Criteria in Solid Tumors (RECIST) will be used to assess the response. It is a standard way to measure how well a cancer patient responds to treatment. It is based on whether tumors shrink, stay the same, or get bigger after there must be at least one tumor that can be measured by CT scans, MRI scans, or PET scan (every 8-12 weeks)where "Complete response" (CR) defined as the disappearance of all tumor lesions, "partial response" (PR) as a reduction of > 30% and they will be stable disease" (SD) as a reduction of < 30% or a growth of < 20% and "progressive disease" (PD) as growth of > 20% or the occurrence of new lesions; all changes will be relative to the baseline imaging. Non-responders are patients with stable disease (SD) or progressive disease (PD). Patients will be separated into three groups:

1. The first group is the responder (Complete response and partial response)
2. The second group is the no responder (progressive disease and stable disease) To explore the association between SNPs and BEV treatments, we will explore the association of VEGFA polymorphisms with BEV's therapeutic efficacy in CRC patients. ORR, DCR, and PFS will estimate the results.

ORR is the Objective response rate Percentage of patients whose disease decreased (Partial response - PR) and/or disappeared (Complete response - CR) after treatment. Disease Control Rate (DCR) is defined as the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response, and stable disease to therapeutic intervention in clinical trials of anticancer agents, and PFS (progression-free survival is defined as the interval from the date on which treatment with bevacizumab was initiated to tumor progression)

ELIGIBILITY:
Inclusion Criteria:

* All eligible patients will be age over 18 years old. The risk of colorectal cancer increases with age; 90% of cases are diagnosed in individuals 50 years of age and older.
* Most patients had a performance status (WHO = 0-2), which is a score that estimates the patient's ability to perform certain activities of daily living (ADLs) without the help of others. Performance status (PS) is one of the strongest prognostic factors for survival in metastatic colorectal cancer patients.
* In all cases, the initial tumor site will be the colon.
* Adult patients already diagnosed with metastatic CRC and received bevacizumab and chemotherapy consisting of fluorouracil and leucovorin or capecitabine in combination with either oxaliplatin (FOLFOX or XELOX) or irinotecan (FOLFIRI or XELIRI).
* Chronic disease patients will be involved

Exclusion Criteria:

* Patient received bevacizumab and chemotherapy for inadequate cycles; the adequate cycle should be not less than three cycle
* Patients participating in the study and not receive bevacizumab owing to risk factors for serious adverse events like GI perforation, Wounds that don't heal, Serious bleeding, Severe high blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Complete response rate (CR) | At the end of Cycle 3 (each cycle is 21 days)
  Every target lesion disappears. Any troublesome lymph nodes, whether they are target or non-target, need to have at least 10 mm removed from their short axis
Partial Response rate (PR) | At the end of Cycle 3 (each cycle is 21 days)
  No less than of 30% reduction in the intended lesion sum diameters, using use the baseline sum diameters as a guide
Progressive Disease rate (PD) | At the end of Cycle 3 (each cycle is 21 days)
  Target lesions' total diameters should rise by at least 20%, applying the smallest overall diameters serving as a guide. (Note: the emergence of one or more additional lesions is likewise regarded as progression)
Stable Disease rate (SD) | At the end of Cycle 3 (each cycle is 21 days)
  There is neither enough rise nor enough reduction to be acceptable as PR or PD, using the lowest total diameters as a reference
Overall survival (OS) | At the end of Cycle 3 (each cycle is 21 days)
  The duration by months from chance to death for all patients who received Bevacizumab was calculated additionally, we excluded any patients who were still alive or lost to follow-up at the time of assessment
Progression free survival (PFS) | At the end of Cycle 3 (each cycle is 21 days)
  The number of months, for all patients alive at the time of assessment from selection of patients until the first sign of disease advancement or death
Objective Response Rate (ORR) | At the end of Cycle 3 (each cycle is 21 days)
  It is the proportion of participants in a therapy group that, within a particular period of time, respond completely or partially to the treatment
Disease control rate (DCR) | At the end of Cycle 3 (each cycle is 21 days)
  The percent (%) of patients with advanced cancer who have seen a full response, only partial response, or stable illness as a result of their therapeutic intervention

SECONDARY OUTCOMES:
Health related quality of life measure (HRQL) | At the end of Cycle 3 (each cycle is 21 days)
  It is a crucial measure that shows clinical benefit and is patient-reported. It is an assessment of a patient's QOL in relation to their health over an extended period of time. The QLQ-C30 version 3.0 tool, developed by the "European -Organization -for Research and Treatment of Cancer" (EORTC), is used to evaluate how colorectal cancer affects a person's QOL. This survey was approved straight from the EORTC Data Centre in Belgium after it was translated and verified in a number of languages, including Arabic language.
Adverse effects (AE) rate | At the end of Cycle 3 (each cycle is 21 days)
  Asessment of any AE that occur during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Baghdad Medical city, Baghdad, Iraq